CLINICAL TRIAL: NCT00344812
Title: Opioid Maintenance Medications Comparison Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPR-95-07-24-03
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-03

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone

INTERVENTIONS:
Drug: LAAM. buprenorphine and methadone

SUMMARY:
A 17 week, double-blind, randomized, parallel group, four arm design outpatient study comparing LAAM, buprenorphine and two dose levels of methadone for the treatment of opioid dependence.

ELIGIBILITY:
Inclusion

* age 21 to 55 years
* diagnosis of opioid dependence by criteria of the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
* evidence of recent opioid use on toxicologic screening

Exclusion

* serious medical or psychiatric illness requiring long-term medication
* positive pregnancy test

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220
Dates: Start 1996-01; Study Completion 1998-06

PRIMARY OUTCOMES:
Study retention
Drug use

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Rolley E Johnson, PharmD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit; Johns Hopkins Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Result] Johnson RE, Chutuape MA, Strain EC, Walsh SL, Stitzer ML, Bigelow GE. A comparison of levomethadyl acetate, buprenorphine, and methadone for opioid dependence. N Engl J Med. 2000 Nov 2;343(18):1290-7. doi: 10.1056/NEJM200011023431802. PMID 11058673